CLINICAL TRIAL: NCT05897801
Title: A CLINICAL STUDY OF THE MeMed BV® TEST TO DISTINGUISH BETWEEN BACTERIAL AND VIRAL INFECTIONS AND LIMIT GUT COLONIZATION BY MULTIDRUG RESISTANT MICROORGANISMS
Brief Title: Distinguishing Bacterial and Viral Infections by MeMed BV® Test to Limit Gut Colonization by MDRO
Acronym: CRONUS
Status: Completed | Type: Observational
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Other Study IDs: CRONUS
Record Dates: First submitted 2023-05-22; First posted 2023-06-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Viral Infection; Bacterial Infections; Multi-antibiotic Resistance; Respiratory Tract Infections
Keywords: Infections; Gut colonization; Respiratory track infections
MeSH Terms: conditions — Virus Diseases; Bacterial Infections; Respiratory Tract Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a respiratory tract infection: Patients entering the emergency department of the sites, presenting with symptoms compatible with the diagnosis of respiratory tract infection.
  Interventions: Diagnostic Test: MeMed BV®

INTERVENTIONS:
Diagnostic Test: MeMed BV® — One blood sampling of 3ml will be drawn on the first day for the performance of the MeMed BV® test. Two rectal swabs will be taken for determining the MDRO gut colonization. Patient information regarding the specific respiratory tract infection and the treatment regimen being prescribed will be recorded in the eCRF made specifically for this trial.

SUMMARY:
The fast increase of Multidrug-resistant microorganisms (MDRO) due to the high amount of antimicrobials being poorly used may be limited by better regulating antimicrobial usage globally. The goal of this observational study is the performance of the MeMed BV® test in the MeMed Key® device at the emergency department to a) support the differential diagnosis between bacterial and viral infections of the respiratory tract and b) provide evidence of how the use of this test may limit gut colonization by MDRO.

DETAILED DESCRIPTION:
Antimicrobial resistance is one of the major threats to the society. One major driver of this phenomenon is the extensive use of antibiotics particularly during the winter months as empirical use for respiratory tract infections. Most of these infections, namely acute exacerbation of chronic obstructive pulmonary disease (AECOPD) and acute bronchitis, are of viral origin and no antibiotics need to be prescribed. To limit the ambiguity of prescribing physicians leading them to unnecessary prescription of antibiotics, one new point-of-care test has been developed which may assist to distinguish between bacterial and viral infections.

This test is called MeMed BV® and is providing the integrative information of three measurable parameters in blood, namely TRAIL (tumour necrosis factor-related apoptosis-inducing ligand), IP-10 (interferon-gamma-induced protein-10) and CRP (C-reactive protein). TRAIL and CRP are increased in the case of bacterial infection; IP-10 is increased in viral infections; and the integrative algorithm suggests the likelihood for a patient to present with bacterial infection, with viral infection or to be at an intermediate state. Based on the results of the Appolo clinical study, the use of the MeMed BV® test which runs in the MeMed Key® device have been registered by the European Medicines Agency and by the Food and Drug Administration (FDA) of the United States for use in the Emergency department (ED) of differentiate between bacterial and viral infections.

The present study is aiming to the performance of the MeMed BV® test in the MeMed Key® device at the ED to a) support the differential diagnosis between bacterial and viral infections of the respiratory tract and b) provide evidence of how the use of this test may limit gut colonization by MDRO.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Both genders
* Written informed consent provided by participants or their legal representatives
* Symptoms compatible with the diagnosis of respiratory tract infection defined as at least one of: fever (core temperature more than or equal to 37.50C), chills, sore throat, myalgias, sudden onset of headache, running nose
* Onset of symptoms the last 7 days

Exclusion Criteria:

* Fever (core temperature more than or equal to 37.50C) for more than 7 days
* Neutropenia defined as less than 1,000 neutrophils/mm3
* Intake of chemotherapy for any malignancy
* Intake of radiotherapy for any malignancy
* Medical history of known active infection by the human immunodeficiency virus (HIV) or hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Pregnancy or lactation
* Any acute trauma
* Any operation the last 7 days
* Presence of acute burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening will be done for the inclusion and exclusion criteria in all patients admitted in the participating sites. Participants will be patients meeting all inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The change of the physicians decisions for the prescribed treatment based on the MeMed BV® test | Through study completion, an average of 1 year
  The change of the physicians decisions for the prescribed treatment based on the MeMed BV® test

SECONDARY OUTCOMES:
The accurate prediction of the viral or the bacterial infection a patient is suffering from using the MeMed BV® test | Through study completion, an average of 1 year
  The accurate prediction of the viral or the bacterial infection a patient is suffering from using the MeMed BV® test
Exploratory endpoint | Through study completion, an average of 1 year
  The rate of gut colonization by MDRO between patients for whom physician decision to receive antibiotics was impacted by the results of the MeMed BV® test and patients for whom physician decision to receive antibiotics was not impacted by the results of the MeMed BV®.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD,PhD, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (3):
- Greece (3):
  - Emergency Department of ATTIKON University General Hospital, Attiki, Chaidari
  - Emergency Department of Tzaneion General Hospital, Attiki, Piraeus
  - General Hospital of Elefsina 1st Department of Internal Medicine, Elefsina

IPD SHARING:
Plan to Share IPD: No